CLINICAL TRIAL: NCT03182842
Title: Evaluation of FreeStyle Libre Flash Glucose Monitoring System During a Children With Type 1 Diabetes Summer Camp - The Free Summer Study
Brief Title: FreeStyle Libre FGM During Summer Camp for Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Free-Summer-01
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FreeStyle Libre FGM (Experimental): Insulin dosing based on FreeStyle Libre FGM glucose values
  Interventions: Device: FreeStyle Libre FGM
- SMBG - Blinded Sensor - Control (Active Comparator): Insulin dosing based on SMBG, FreeStyle Libre FGM will be blinded.
  Interventions: Device: SMBG - Blinded Sensor

INTERVENTIONS:
Device: FreeStyle Libre FGM — Insulin dosing based on FreeStyle Libre FGM system that is indicated for measuring interstitial fluid glucose levels in people (age 4 and older) with diabetes mellitus.
  Other Names: Intervention - Sensor ON
  Arms: FreeStyle Libre FGM
Device: SMBG - Blinded Sensor — Insulin dosing based on SMBG
  Other Names: Control
  Arms: SMBG - Blinded Sensor - Control

SUMMARY:
A randomized, double-blinded, single center, parallel design pediatric study, on 45 subjects with type 1 diabetes (T1D), aged six to 15 (inclusive) years, measuring sensor time in glucose values within range 3.9 - 10 mmol/l (70 - 180 mg/dl) achieved using the FreeStyle Libre Flash Glucose Monitoring System (FGM - intervention, Abbott Diabetes Care, California, USA) versus Self-Monitoring Blood Glucose (SMBG - control).

Study duration will be two weeks per subject and two weeks overall, it will take place at youth summer camp for children with T1D. Main inclusion criteria include age of six to 15 (inclusive) years, clinical diagnosis of T1D for at least six months, at least three months of current use of insulin pump therapy, HbA1c between 6.3 and 10 % (both inclusive), no other chronic medical conditions (beside treated hypothyroidism and celiac disease) and no current medications (other than insulin) (detailed list of inclusion and exclusion criteria list can be found at section 6).

The objectives of this clinical investigation is:

1. to evaluate the efficacy of glucose control using the FreeStyle Libre FGM in children with T1D during two weeks of summer camp.

ELIGIBILITY:
Inclusion Criteria:

- 1. The subject has documented T1D, as defined by the American Diabetes Association and World Health Organization (ADA/WHO) for at least six month prior to study enrolment 2. Documented evidence should exist within the patient history of T1D 3. The subject is between six and 15 years of age (inclusive) at the time of enrolment 4. The subject has been treated with an insulin pump for at least 3 months 5. The subject has an A1C value between 6.3 and 10% (both inclusive) based on analysis from the local laboratory. A1C testing must follow National Glycohemoglobin Standardization Program (NGSP) standards.

6. The subject is willing to follow all study instructions 7. Subject is willing to perform daily self-monitoring of blood glucose (SMBG). 8. If subject has celiac/Hashimoto disease, the disease has to be adequately treated as determined by the investigator 9. Subject has a BMI above 5th centile and below 95th centile for age, respectively.

Exclusion Criteria:

* 1. Concomitant diseases that influence metabolic control (e.g. anemia, significantly impaired hepatic function, renal failure, history of adrenal insufficiency) or other medical conditions, which in the investigator's opinion, may compromise patient safety; Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment.

  2. Significant co-morbidity that, in the opinion of the investigators would preclude participation in the study (e.g. current treatment for cancer, mental disorder) 3. Subject is taking or has taken oral or parenteral glucocorticoids within 1 month prior to screening, or plans to take oral or parenteral glucocorticoids during the study.

  4. Subject is taking antidiabetic agents or other medications, which could be a contraindication to participation in the study by the judgment of the investigator.

  5. Subject is participating in another study of a medical device or drug that could affect glucose measurements or glucose management or Receipt of any investigational medical product within 1 month prior to screening.

  6. Female subject of child-bearing potential who is pregnant, breast-feeding, or planning to become pregnant during the study.

  7. Subject has known hypoglycemic unawareness or recurrent severe hypoglycemic events with seizure and/or coma (more than two episodes) within 6 months prior to screening.

  8. Subject has a history of one or more episodes of Diabetic Ketoacidosis (DKA) requiring hospitalization within a month prior to the screening.

  9. Subject has current or recent history of alcohol or drug abuse. 10. Subject has visual impairment or hearing loss, which in the investigator's opinion, may compromise patient ability to perform study procedures safely (child and parent should be evaluated as a unit).

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Time within 3.9 and 10 mmol/l | Two weeks
  between-group difference (FGM versus SMBG) in time within range of glucose values within 3.9 - 10 mmol/l (70-180 mg/dl) during two weeks of diabetes summer camp based on sensor glucose readings

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, Prof., Principal Investigator — Head, Chair of Pediatrics, Faculty of Medicine Vice Dean for Research, Faculty of Medicine
Locations (1):
- Medical Faculty - University of Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Piona C, Dovc K, Mutlu GY, Grad K, Gregorc P, Battelino T, Bratina N. Non-adjunctive flash glucose monitoring system use during summer-camp in children with type 1 diabetes: The free-summer study. Pediatr Diabetes. 2018 Nov;19(7):1285-1293. doi: 10.1111/pedi.12729. Epub 2018 Aug 16. PMID 30022571